CLINICAL TRIAL: NCT05042180
Title: Virtual Reality-Assisted Cognitive Behavioral Therapy for Alcohol Dependence: A Randomized Controlled Trial (CRAVR)
Brief Title: Virtual Reality-Assisted Cognitive Behavioral Therapy for Alcohol Dependence (CRAVR)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Psychiatric Centre Rigshospitalet (Other)
Collaborators: The Novavì outpatient clinics, Copenhagen (Unknown)
Responsible Party: Principal Investigator, Anders Fink-Jensen, MD, DMSci, Professor, MD, DMSci, Psychiatric Centre Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRAVR
Record Dates: First submitted 2021-07-27; First posted 2021-09-13 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Alcohol Dependence, in Remission; Addiction, Alcohol
Keywords: Alcohol; Addiction; Virtual Reality; Exposure Therapy; Cognitive Behavioral Therapy
MeSH Terms: conditions — Alcoholism; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: single-blinded, randomized, controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Cognitive Behavioral Therapy (VRCBT) (Experimental): The VR exposure is performed to induce alcohol craving and high-risk induced reactions during the therapy session, in order to trigger a lifelike response to alcohol, while the therapist is present and able to train the participant in applying CBT-based coping strategies to deal with the alcohol cravings.
  Interventions: Behavioral: Virtual Reality Cognitive Behavioral Therapy (CRAVR)
- Cognitive Behavioral Therapy (CBT) (Active Comparator): CBT is made up of the following elements: i) recognition (ii) avoiding and (iii) overcoming drinking cravings in high-risk situations with the aim of preventing relapse.
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: Virtual Reality Cognitive Behavioral Therapy (CRAVR) — Participants in the intervention group will scheduled for 14 treatment sessions based on manualized cognitive behavioral therapy assisted with alcohol-related high risk situations in virtual reality. VR-assisted gradual exposure therapy is integrated as a part of CBT. I.e. VR scenes are used in CBT to induce craving for coping strategy skill training and cognitive analysis.
  Arms: Virtual Reality Cognitive Behavioral Therapy (VRCBT)
Behavioral: CBT — The active comparator receives 14 conventional cognitive behavioral therapy sessions with
  Arms: Cognitive Behavioral Therapy (CBT)

SUMMARY:
The study is a single-blinded, randomized, controlled, 12 months clinical trial. The objective is to investigate the feasibility, effects and side-effects of virtual reality-assisted cognitive behavioral therapy (VR-CBT) vs. cognitive behavioral therapy (CBT) in patients with a diagnosis of alcohol dependence.

DETAILED DESCRIPTION:
Recruitment of participants:

102 patients will be recruited from the Novaví outpatient clinics, where they will be informed orally and in writing about the research project and, if they are interested, an information meeting is booked. If patients show symptoms of abstinence, these are treated prior to the information meeting by doctors and nurses in Novaví. If the patient then wishes to participate and meets the inclusion criteria, informed consent is obtained and screening is performed using the questionnaires described later. Included patients will then be randomized to either:

1. Virtual reality-assisted cognitive behavioral therapy (VR-CBT)
2. Cognitive behavioral therapy (CBT) without VR (control group)

Screening:

At the screening sessions, patients' medical history is obtained, as well as their alcohol intake over the past 30 days recorded via Timeline Follow-Back (TLFB). Patients are also asked about previous alcohol dependence treatment and general information about psychosocial factors incl. education, work, marital status, and functional level using Global Assessment of functioning (GAF). In addition, alcohol-related problems are assessed using the Alcohol Users Identification Test (AUDIT), abstinence using the Clinical Institute Withdrawal Assessment of Alcohol Scale Revised (CIWA-Ar), intake of other drugs using the Drug User Identification Test (DUDIT), and alcohol craving using the Penn Alcohol Craving Scale (PACS). The Becks questionnaires, Depression Inventory 2 (BDI-II) and Beck's Anxiety Inventory (BAI), are included to assess the degree of anxiety and depression, and in addition, tests of mental function are performed using the Screening for Cognitive Impairment in Psychiatry (SCIP).

Intervention:

Included participants will in collaboration with their therapist schedule a standard course of treatment based on national guidelines from health authorities. After inclusion, participants are randomized to either:

1. 14 sessions of VR-CBT (Group A)
2. 14 sessions of CBT without VR (Group B, control group)

The participants in group A are exposed to VR-simulated high-risk situations filmed in a restaurant, a pub, at home, at a party or at the supermarket, to trigger alcohol cravings and other high-risk induced reactions of which the participants are subsequently trained to handle by trained therapists using CBT-based techniques.

The participants in group B receive the same treatment without VR exposure. The will be 4 weeks of weekly-biweekly treatment, followed by 20-21 weeks of treatment every 2-3 weeks, which is in line with the standard treatment in the Novaví outpatient clinics. The intervention deviates from standard treatment, as none of the participants receive pharmaceutical alcohol treatment during the treatment period (6 months) except for abstinence treatment if needed.

Randomization and blinding:

After screening a patient (ensuring that all inclusion criteria and no exclusion criteria are met) the patient is included. Participants are randomly allocated to either VR-CBT og CBT, 51 participants in each group. Randomization takes place in REDCap, which is a secure web application for building and managing surveys and databases. Age, sex and alcohol consumption are stratified at the time of inclusion ('heavy drinking days' and alcohol consumption - evaluated by TLFB). The technical setup of the randomization tool is performed in close collaboration with an expert in statistics, which ensures correct functionality before starting the experiment. After randomization, the therapist ensures that the participant receives the correct treatment and performs the alcohol craving assessment during each VR-CBT session unblinded using visual analog score (VAS). The study staff conducting the remaining data collections and the entire data analysis remain blinded until the database is opened at the end of the study. In situations where it is necessary to break the blind, it is possible to change the user rights in REDCap and gain access to the randomization tools. With the randomization tools, it is possible to detect the treatment (VR-CBT or CBT) based on study ID and all activities performed in REDCap are registered in the program.

Follow-up:

Each participant must attend a follow-up visit 3, 6, and 12 months from inclusion, where data collection will take place using the before mentioned questionnaires. The follow-up visit will be approx. 1 hour.

Statistical analysis:

All statistical analyzes are performed using the intention-to-treat principle, where all patients who have become randomized and has received a minimum of 1 session of VR-CBT (group A) or CBT without VR (group B), is included in the analysis. Missing data are implemented through the multiple imputation method and the analyzes are performed in the program "R" with alpha = 0.05 and 2-sided test. All continuous effect measures are analyzed using ANOVA from baseline to most recent measurement, and categorical data are analyzed using chi2 analysis. All data distributions will be assessed for normality by visual inspection of histogram and by Q-Q plots. If data is not normally distributed, log transformation is performed, and if this is not successful, non-parametric testing is used.

ELIGIBILITY:
Inclusion Criteria:

* Informed oral and written consent
* Meets criteria for alcohol dependence syndrome according to International Classification of Diseases (ICD) 10, WHO & Diagnostic and Statistical Manual of Mental Disorder (DSM-5)
* Age 18 - 70 years old (both included)
* Minimum 5 'heavy drinking days' in the last month, which is defined as an alcohol intake above 60/48 grams or 5/4 items per. day for resp. men and women over the past 30 days

Exclusion Criteria:

* Other active substance use defined by DUDIT score> 6 (for men)> 2 (for women) and meet the criteria for other drug dependence according to ICD-10 (excluding nicotine)
* Does not speak or understand Danish
* Mental retardation or known severe psychiatric illness or other condition where it is assessed that will interfere with participation eg severely impaired vision or hearing.
* Medical alcohol treatment (disulfiram, acamprosate, naltrexone or nalmefen) within the latest 4 weeks and during the treatment period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in total alcohol consumption | Baseline, 6 months, 9 months, 12 months
  Percent change in alcohol consumption, defined as "x" grams of alcohol for past 30 days. This will be registered using the Timeline-Follow-Back (TLFB) method.

SECONDARY OUTCOMES:
Change in heavy drinking days | Baseline, 6 months, 9 months, 12 months
  Based on the past 30 days of alcohol consumption using time line follow-back (TLFB), heavy drinking days are evaluated. 1 heavy drinking day consists of alcohol consumption exceeding 60/48 grams for men and women respectively.
Change in Alcohol Users Identification Test (AUDIT) score | Baseline, 6 months, 9 months, 12 months
  Screening for excessive drinking. Higher score = worse outcome
Change in Drug User Identification Test (DUDIT) score | Baseline, 6 months, 9 months, 12 months
  Identification of individuals with drug-related problems. Higher score = worse outcome
Change in Penn Alcohol Craving Scale (PACS) score | Baseline, 6 months, 9 months, 12 months
  Assessing alcohol craving. Higher score = worse outcome
Screening for Cognitive Impairment in Psychiatry (SCIP) score | Baseline, 6 months, 9 months, 12 months
  The 20 minute test is a scale developed for screening cognitive deficits. Higher score = better outcome
Change in Global Assessment of functioning (GAF) score | Baseline, 6 months, 9 months, 12 months
  GAF measures to what degree a person's symptoms affect their daily functioning on a scale of 0 to 100. Higher score = better outcome
Becks Anxiety Inventory (BAI) score | Baseline, 6 months, 9 months, 12 months
  Measures the severity of anxiety. Higher score = worse outcome
Becks Depression Inventory 2 (BDI-II) score | Baseline, 6 months, 9 months, 12 months
  Measures the severity of depression. Higher score = worse outcome
Simulator Sickness Questionnaire (SSQ) | Each of the 14 treatment sessions over 6 months
  Measures whether participants experience symptoms of simulator sickness while in Virtual Reality. Higher score = worse outcome
VR-induced craving on a visual analog scale (VAS) | Each of the 14 treatment sessions over 6 months
  For each of the 6 VR-scenes, craving is evaluated before, during and after exposure as well as at the end of the therapy session
Alcohol withdrawal symptoms | Evaluated at inclusion
  Alcohol withdrawal symptoms are evaluated at inclusion. Higher score = worse outcome
Qualitative assessment | After completion of a full treatment period of 6 months
  15 patients and 5 therapists will be asked about advantages and disadvantages of using virtual reality

CONTACTS AND LOCATIONS:
Locations (1):
- Novavi ambulatorierne, Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thaysen-Petersen D, Hammerum SK, Vissing AC, Oestrich IH, Nordentoft M, During SW, Fink-Jensen A. Virtual reality-assisted cognitive behavioral therapy for patients with alcohol use disorder: a randomized feasibility study. Front Psychiatry. 2024 Feb 14;15:1337898. doi: 10.3389/fpsyt.2024.1337898. eCollection 2024. PMID 38419905
- [Derived] Thaysen-Petersen D, Hammerum SK, Vissing AC, Arnfred BT, Nordahl R, Adjorlu A, Nordentoft M, Oestrich IH, During SW, Fink-Jensen A. Virtual reality-assisted cognitive behavioural therapy for outpatients with alcohol use disorder (CRAVR): a protocol for a randomised controlled trial. BMJ Open. 2023 Mar 29;13(3):e068658. doi: 10.1136/bmjopen-2022-068658. PMID 36990475